CLINICAL TRIAL: NCT02218697
Title: Immunogenicity and Safety Study of GSK Biologicals' Quadrivalent Split Virion Influenza Vaccine 2014/2015 Influsplit™ Tetra (Fluarix™ Tetra) (GSK2321138A) When Co-administered With Pneumovax™ 23 in Adults 50 Years of Age and Older
Brief Title: Evaluation of the Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Quadrivalent Influenza Vaccine Influsplit™ Tetra (Fluarix™ Tetra) (GSK2321138A) When Co-administered With Pneumovax™ 23 in Adults 50 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 117276; 2014-001118-24 (EudraCT Number)
Record Dates: First submitted 2014-08-14; First posted 2014-08-18 (Estimated); Results first posted 2017-03-09 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Influenza
Keywords: Immunogenicity; Influsplit Tetra (Fluarix Tetra) 2014/2015 season; Safety; Adults; Pneumovax 23/Pneumovax; Co-administration; Elderly; Seasonal influenza; Pneumococcal infection
MeSH Terms: conditions — Influenza, Human; Pneumococcal Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-Ad Group (Experimental): Subjects received 1 dose of Influsplit™ Tetra vaccine and 1 dose of Pneumovax™ 23 vaccine at Day 0 and 1 dose of placebo at Day 28.
  Interventions: Biological: Influsplit™ Tetra (Fluarix™ Tetra); Biological: Pneumovax™ 23; Biological: Placebo (Saline)
- Control Group (Experimental): Subjects received 1 dose of Influsplit™ Tetra vaccine and 1 dose of placebo at Day 0 and 1 dose of Pneumovax™ 23 vaccine at Day 28.
  Interventions: Biological: Influsplit™ Tetra (Fluarix™ Tetra); Biological: Pneumovax™ 23; Biological: Placebo (Saline)

INTERVENTIONS:
Biological: Influsplit™ Tetra (Fluarix™ Tetra) — Intramuscular injection, 1 dose each in Control and Co-Ad groups.
  Other Names: D-QIV; GSK2321138A
Biological: Pneumovax™ 23 — Intramuscular injection, 1 dose each in Control and Co-Ad groups.
Biological: Placebo (Saline) — Intramuscular injection, 1 dose each in Control and Co-Ad groups.

SUMMARY:
The purpose of this study is to investigate the immunogenicity and safety when GSK Biologicals' influenza vaccine Influsplit™ Tetra (Fluarix™ Tetra) is co-administered with Merck & Co. Inc.'s pneumococcal vaccine (Pneumovax™23/Pneumovax) in adults 50 years of age and older at risk for complications from influenza and pneumococcal infections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits).
* A male or female aged 50 years or above at the time of the first vaccination at risk for complications from influenza and/or pneumococcal infections, meeting their respective countries' recommendations for vaccination against influenza and pneumococcal disease.

  * At risk subjects include adults with chronic respiratory, heart, kidney, liver or neurological disease; human immunodeficiency virus (HIV) disease on combination antiretroviral therapy (cART) with cluster of differentiation 4 (CD4) T-cell counts greater than 350 cells/mm3; sickle cell disease or coeliac syndrome that may lead to splenic dysfunction (all other asplenics are excluded). The decision to enrol should be based on the investigators clinical judgement.
* Written informed consent obtained from the subject.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. Inhaled, topical and low-dose intra-articular steroids are allowed.
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before the first dose and 30 days after the last dose of vaccine.
* Administration of such a vaccine has to be documented in the "Concomitant vaccination" of the electronic Case Report Form (eCRF).
* Administration of long-acting immune-modifying drugs/treatment within six months prior to the first vaccine dose or expected administration at any time during the study period. These immunosuppressant drugs/treatment/Biologics include:

  * Methotrexate
  * Leflunomide
  * Azathioprine and 6-mercaptopurine
  * Cyclosporin A
  * Cyclophosphamide
  * Tacrolimus, everolimus, sirolimus, temsirolimus
  * Mycophenolate mofetil
  * Antilymfocytaire immunoglobulins
  * Tumor Necrosis Factor (TNF) inhibitors: Adalimumab (Humira®), certolizumab (Cimzia®), etanercept (Enbrel®), golimumab (Simponi®) and infliximab(Remicade®)
  * Monoclonal antibodies and other biologicals: Rituximab (Mabthera®), Abatacept (Orencia®), tocilizumab (RoActemra®), basiliximab (Simulect®), Natalizumab (Tysabri®) cluster of differentiation 3 (CD3), …
  * Antitumor agents: alkylating agents, antimetabolites, antitumor antibiotics, topoisomerase inhibitors, microtubule inhibitors and other anti-tumor agents
  * Lenalidomide Revlimid®
  * Tasonermin: Beromun®
  * Proleukin® (aldesleukin; Novartis, …)
  * Tyrosine kinase inhibitor (Glivec®)Omalizumab Xolair®
  * Eculizumab Soliris® The above list is compiled from: [Federal Public Service Belgium: Health, Food Chain Safety and Environment].
  * Any immunosuppressive treatment which in the opinion of the investigator will not allow an adequate immune response. Inhaled, topical and low-dose intra-articular steroids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination with a pneumococcal vaccine within the last five years.
* Previous vaccination with an influenza vaccine within the last six months.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination. HIV infected subjects on cART with CD4 T-cell counts above 350 cells/mm3 can be enrolled.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥ 38.0°C (100.4°F). The preferred route for recording temperature in this study will be axillary.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever [≥ 38.0°C (100.4°F)] may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study or would make intramuscular (IM) injection unsafe.
* Asplenia or dysfunction of the spleen. This excludes homozygous sickle cell disease or coeliac syndrome that may lead to splenic dysfunction.
* Acute clinically significant (i.e. a medically significant change from baseline condition in the past 30 days) pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* History of chronic alcohol consumption and/or drug abuse.
* History of Guillain-Barré syndrome.
* A history of anaphylaxis following ANY vaccination.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-01-14 (Actual); Study Completion 2015-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, Ghent, Belgium
- France (5):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Laval
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Saint-Cyr-sur-Loire
  - GSK Investigational Site, Tours

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Ofori-Anyinam O, Leroux-Roels G, Drame M, Aerssens A, Maes C, Amanullah A, Schuind A, Li P, Jain VK, Innis BL. Immunogenicity and safety of an inactivated quadrivalent influenza vaccine co-administered with a 23-valent pneumococcal polysaccharide vaccine versus separate administration, in adults >/=50years of age: Results from a phase III, randomized, non-inferiority trial. Vaccine. 2017 Nov 1;35(46):6321-6328. doi: 10.1016/j.vaccine.2017.09.012. Epub 2017 Oct 5. PMID 28987445
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 117276 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 117276 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 117276 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 117276 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 117276 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 117276 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 117276 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the Control Group, 2 subjects withdrew at Day 0. In the Co-Ad Group, 4 subjects withdrew at Day 0, 1 subject withdrew at Day 28 and 1 subject withdrew at Day 56.
Pre-assignment Details: Of the 357 subjects enrolled, 1 subject failed to meet the inclusion criteria hence he/she was excluded from study start.
Period: Overall Study
Arm/Group | Control Group | Co-Ad Group
Started | 179 | 177
Completed | 177 | 171
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Unwilling to be vaccinated in left arm | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Co-Ad Group | Total
Number analyzed (Participants) | 179 | 177 | 356
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (9.4) | 68.1 (9.0) | 68.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 76 | 153
  Male | 102 | 101 | 203
Race/Ethnicity, Customized [Number; unit: Participants]
  African Heritage / African American | 1 | 2 | 3
  White - Arabic / North African Heritage | 3 | 1 | 4
  White - Caucasian / European Heritage | 175 | 172 | 347
  Mixed Origin | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies Titers Against the 4 Vaccine Strains.
Description: HI antibody titres were expressed as geometric mean titers (GMTs) and adjusted GMT ratios (Control Group/Co-Ad Group). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), FluA/Texas/50/2012 (H3N2), Flu B/Brisbane/60/2008 (Victoria) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 28 post Influsplit™ Tetra vaccination
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects who received the study vaccine according to their treatment assignment and for whom the assay results for antibodies against at least one study vaccine strain after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 170 | 163
Titers
  H1N1 | 253.2 [205.3 to 312.1] | 235.5 [195.0 to 284.5]
  H3N2 | 73.6 [62.1 to 87.1] | 78.6 [65.2 to 94.7]
  Victoria | 178.7 [154.9 to 206.2] | 157.9 [136.4 to 182.9]
  Yamagata | 346.5 [302.3 to 397.1] | 353.8 [310.5 to 403.2]
Statistical Analysis 1: Comparison: Control Group vs Co-Ad Group; The adjusted GMT of HI antibodies for H1N1 strain at Day 28 post Influsplit™ Tetra vaccination, the GMT ratio of Control group/Co-Ad group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination titer as covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion (for each of the 4 strains): UL of the 95% CI for the GMT ratio (Control Group / Co-Ad Group) does not exceed 2.0; ANCOVA; Adjusted GMT ratio = 1.13, 95% CI 2-sided [0.88 to 1.46] — The GMTs were used to calculate the Adjusted GMTs, which in turn were used to calculate the Adjusted GMT ratio with 95% confidence interval
Statistical Analysis 2: Comparison: Control Group vs Co-Ad Group; The adjusted GMT of HI antibodies for H3N2 strain at Day 28 post Influsplit™ Tetra vaccination, the GMT ratio of Control group/Co-Ad group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination titer as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Adjusted GMT ratio = 0.97, 95% CI 2-sided [0.78 to 1.21] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Control Group vs Co-Ad Group; The adjusted GMT of HI antibodies for Victoria strain at Day 28 post Influsplit™ Tetra vaccination, the GMT ratio of Control group/Co-Ad group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination titer as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Adjusted GMT ratio = 1.17, 95% CI 2-sided [0.98 to 1.40] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Control Group vs Co-Ad Group; The adjusted GMT of HI antibodies for Yamagata strain at Day 28 post Influsplit™ Tetra vaccination, the GMT ratio of Control group/Co-Ad group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titers, including the vaccine group as fixed effect and the pre-vaccination titer as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Adjusted GMT ratio = 0.99, 95% CI 2-sided [0.84 to 1.16] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Pneumococcal Vaccine Response in Terms of Anti-pneumococcal Antibody Concentrations Against 6 Pneumococcal Serotypes (1, 3, 4, 7F, 14 and 19A).
Description: Anti-pneumococcal antibody concentrations were expressed as adjusted geometric mean concentrations (GMCs) and adjusted GMC ratio (Control Group/Co-Ad Group).
Time Frame: At 28 days after Pneumovax™ 23 vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ug per ml
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 169 | 162
ug per ml
  Polysaccharide 01 IgG | 5.5 [4.3 to 7.0] | 4.9 [3.9 to 6.2]
  Polysaccharide 03 IgG | 1.7 [1.4 to 2.1] | 1.7 [1.4 to 2.0]
  Polysaccharide 04 IgG: number analyzed (Participants) | 169 | 161
  Polysaccharide 04 IgG | 2.3 [1.8 to 2.9] | 1.7 [1.4 to 2.2]
  Polysaccharide 7F IgG | 9.0 [6.9 to 11.8] | 8.1 [6.2 to 10.6]
  Polysaccharide 14 IgG | 20.2 [16.0 to 25.6] | 14.1 [11.3 to 17.6]
  Polysaccharide 19A IgG | 9.2 [7.1 to 11.9] | 7.7 [6.1 to 9.8]
Statistical Analysis 1: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody concentrations for Polysaccharide 01 serotype at Day 28 post Pneumovax™ 23 vaccination, the GMC ratio of Control Group/Co-Ad Group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titres/concentrations, including the vaccine group as fixed effect and the pre-vaccination titre/concentration as covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion (for each of six pneumococcal serotypes): UL of the 95% CI for the geometric mean concentration (GMC) ratio (Control group over Co-Ad group) does not exceed 2.0; ANCOVA; Adjusted GMC ratio = 1.14, 95% CI 2-sided [0.86 to 1.50] — The GMCs were used to calculate the Adjusted GMCs, which in turn were used to calculate the Adjusted GMC ratio with 95% confidence interval
Statistical Analysis 2: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody concentrations for Polysaccharide 03 serotype at Day 28 post Pneumovax™ 23 vaccination, the GMC ratio of Control Group/Co-Ad Group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titres/concentrations, including the vaccine group as fixed effect and the pre-vaccination titre/concentration as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMC ratio = 1.18, 95% CI 2-sided [0.96 to 1.45] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody concentrations for Polysaccharide 04 serotype at Day 28 post Pneumovax™ 23 vaccination, the GMC ratio of Control Group/Co-Ad Group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titres/concentrations, including the vaccine group as fixed effect and the pre-vaccination titre/concentration as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMC ratio = 1.26, 95% CI 2-sided [0.98 to 1.62] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody concentrations for Polysaccharide 7F serotype at Day 28 post Pneumovax™ 23 vaccination, the GMC ratio of Control Group/Co-Ad Group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titres/concentrations, including the vaccine group as fixed effect and the pre-vaccination titre/concentration as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMC ratio = 1.24, 95% CI 2-sided [0.95 to 1.63] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody concentrations for Polysaccharide 14 serotype at Day 28 post Pneumovax™ 23 vaccination, the GMC ratio of Control Group/Co-Ad Group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titres/concentrations, including the vaccine group as fixed effect and the pre-vaccination titre/concentration as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMC ratio = 1.20, 95% CI 2-sided [0.91 to 1.57] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Control Group vs Co-Ad Group; Anti-pneumococcal antibody concentrations for Polysaccharide 19A serotype at Day 28 post Pneumovax™ 23 vaccination, the GMC ratio of Control Group/Co-Ad Group and the two sided 95% CI were computed by fitting an ANCOVA model on the logarithm10 transformation of the titres/concentrations, including the vaccine group as fixed effect and the pre-vaccination titre/concentration as covariate; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; ANCOVA; Adjusted GMC ratio = 1.34, 95% CI 2-sided [1.05 to 1.70] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Number of Subjects Reporting Solicited Local Adverse Events (AEs)
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain = significant pain at rest and pain that prevented normal everyday activities. Grade 3 redness and swelling = greater than 50 millimeters (mm) i.e. > 100mm.
Time Frame: Within 7 days (Days 0 - 6) after each dose and across doses.
Population: The analysis was performed on the Total Vaccinated cohort which included all subjects with at least one vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 177 | 173
Subjects
  Any Pain, Dose 1 (Influsplit™ Tetra) | 28 | 58
  Grade 3 Pain,Dose 1(Influsplit™ Tetra) | 0 | 2
  Any Pain, Dose 1 (Placebo): number analyzed (Participants) | 176 | 0
  Any Pain, Dose 1 (Placebo) | 10 |
  Grade 3 Pain, Dose 1 (Placebo): number analyzed (Participants) | 176 | 0
  Grade 3 Pain, Dose 1 (Placebo) | 0 |
  Any Pain, Dose 1 (Pneumovax™ 23): number analyzed (Participants) | 0 | 173
  Any Pain, Dose 1 (Pneumovax™ 23) |  | 76
  Grade 3 Pain, Dose 1 (Pneumovax™ 23): number analyzed (Participants) | 0 | 173
  Grade 3 Pain, Dose 1 (Pneumovax™ 23) |  | 6
  Any Redness, Dose 1 (Influsplit™ Tetra) | 3 | 2
  Grade3 Redness,Dose 1(Influsplit™ Tetra) | 0 | 0
  Any Redness, Dose 1 (Placebo): number analyzed (Participants) | 176 | 0
  Any Redness, Dose 1 (Placebo) | 3 |
  Grade 3 Redness, Dose 1 (Placebo): number analyzed (Participants) | 176 | 0
  Grade 3 Redness, Dose 1 (Placebo) | 0 |
  Any Redness, Dose 1 (Pneumovax™ 23): number analyzed (Participants) | 0 | 173
  Any Redness, Dose 1 (Pneumovax™ 23) |  | 8
  Grade 3 Redness, Dose 1 (Pneumovax™ 23): number analyzed (Participants) | 0 | 173
  Grade 3 Redness, Dose 1 (Pneumovax™ 23) |  | 0
  Any Swelling, Dose1 (Influsplit™ Tetra) | 1 | 3
  Grade3 Swelling,Dose1(Influsplit™ Tetra) | 0 | 0
  Any Swelling, Dose 1 (Placebo): number analyzed (Participants) | 176 | 0
  Any Swelling, Dose 1 (Placebo) | 1 |
  Grade 3 Swelling, Dose 1 (Placebo): number analyzed (Participants) | 176 | 0
  Grade 3 Swelling, Dose 1 (Placebo) | 0 |
  Any Swelling, Dose 1 (Pneumovax™ 23): number analyzed (Participants) | 0 | 173
  Any Swelling, Dose 1 (Pneumovax™ 23) |  | 7
  Grade 3 Swelling,Dose 1 (Pneumovax™ 23): number analyzed (Participants) | 0 | 173
  Grade 3 Swelling,Dose 1 (Pneumovax™ 23) |  | 0
  Any Pain, Dose 2 (Influsplit™ Tetra): number analyzed (Participants) | 0 | 0
  Grade 3 Pain, Dose 2 (Influsplit™ Tetra): number analyzed (Participants) | 0 | 0
  Any Pain, Dose 2 (Placebo): number analyzed (Participants) | 0 | 171
  Any Pain, Dose 2 (Placebo) |  | 8
  Grade 3 Pain, Dose 2 (Placebo): number analyzed (Participants) | 0 | 171
  Grade 3 Pain, Dose 2 (Placebo) |  | 0
  Any Pain, Dose 2 (Pneumovax™ 23): number analyzed (Participants) | 177 | 0
  Any Pain, Dose 2 (Pneumovax™ 23) | 63 |
  Grade 3 Pain, Dose 2 (Pneumovax™ 23): number analyzed (Participants) | 177 | 0
  Grade 3 Pain, Dose 2 (Pneumovax™ 23) | 8 |
  Any Redness, Dose 2 (Influsplit™ Tetra): number analyzed (Participants) | 0 | 0
  Grade 3 Redness,Dose 2(Influsplit™ Tetra): number analyzed (Participants) | 0 | 0
  Any Redness, Dose 2 (Placebo): number analyzed (Participants) | 0 | 171
  Any Redness, Dose 2 (Placebo) |  | 1
  Grade 3 Redness, Dose 2 (Placebo): number analyzed (Participants) | 0 | 171
  Grade 3 Redness, Dose 2 (Placebo) |  | 0
  Any Redness, Dose 2 (Pneumovax™ 23): number analyzed (Participants) | 177 | 0
  Any Redness, Dose 2 (Pneumovax™ 23) | 8 |
  Grade 3 Redness, Dose 2 (Pneumovax™ 23): number analyzed (Participants) | 177 | 0
  Grade 3 Redness, Dose 2 (Pneumovax™ 23) | 1 |
  Any Swelling, Dose 2 (Influsplit™ Tetra): number analyzed (Participants) | 0 | 0
  Grade 3 Swelling,Dose 2 (Influsplit™ Tetra): number analyzed (Participants) | 0 | 0
  Any Swelling, Dose 2 (Placebo): number analyzed (Participants) | 0 | 171
  Any Swelling, Dose 2 (Placebo) |  | 0
  Grade 3 Swelling, Dose 2 (Placebo): number analyzed (Participants) | 0 | 171
  Grade 3 Swelling, Dose 2 (Placebo) |  | 0
  Any Swelling, Dose 2 (Pneumovax™ 23): number analyzed (Participants) | 177 | 0
  Any Swelling, Dose 2 (Pneumovax™ 23) | 5 |
  Grade 3 Swelling, Dose 2 (Pneumovax™ 23): number analyzed (Participants) | 177 | 0
  Grade 3 Swelling, Dose 2 (Pneumovax™ 23) | 1 |
  Any Pain, Across Doses (Influsplit™ Tetra) | 28 | 58
  Grade 3 Pain, Across Doses (Influsplit™Tetra) | 0 | 2
  Any Pain, Across Doses (Placebo): number analyzed (Participants) | 176 | 171
  Any Pain, Across Doses (Placebo) | 10 | 8
  Grade 3 Pain, Across Doses (Placebo): number analyzed (Participants) | 176 | 171
  Grade 3 Pain, Across Doses (Placebo) | 0 | 0
  Any Pain, Across Doses (Pneumovax™ 23) | 63 | 76
  Grade 3 Pain, Across Doses (Pneumovax™ 23) | 8 | 6
  Any Redness, Across Doses (Influsplit™Tetra) | 3 | 2
  Grade 3 Redness, Across Doses (Influsplit™ Tetra) | 0 | 0
  Any Redness, Across Doses (Placebo): number analyzed (Participants) | 176 | 171
  Any Redness, Across Doses (Placebo) | 3 | 1
  Grade 3 Redness, Across Doses (Placebo): number analyzed (Participants) | 176 | 171
  Grade 3 Redness, Across Doses (Placebo) | 0 | 0
  Any Redness, Across Doses (Pneumovax™ 23) | 8 | 8
  Grade 3 Redness, Across Doses (Pneumovax™23) | 1 | 0
  Any Swelling, Across Doses (Influsplit™Tetra) | 1 | 3
  Grade 3 Swelling, Across Doses (Influsplit™Tetra) | 0 | 0
  Any Swelling, Across Doses (Placebo): number analyzed (Participants) | 176 | 171
  Any Swelling, Across Doses (Placebo) | 1 | 0
  Grade 3 Swelling, Across Doses (Placebo): number analyzed (Participants) | 176 | 171
  Grade 3 Swelling, Across Doses (Placebo) | 0 | 0
  Any Swelling, Across Doses (Pneumovax™23) | 5 | 7
  Grade 3 Swelling, Across Doses (Pneumovax™23) | 1 | 0

4. Secondary Outcome: Number of Subjects Reporting Solicited General Adverse Events (AEs)
Description: Solicited general symptoms assessed were fatigue, gastrointestinal symptoms*, headache, joint pain, muscle aches, shivering, sweating and fever. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Grade 3 was defined as symptoms that prevented normal everyday activities. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 fever was defined as temperature greater than (>)39.0°C.
  *Gastrointestinal (GI) symptoms included nausea, vomiting, diarrhoea and/or abdominal pain
Time Frame: Within 7 days (Days 0 - 6) after each dose and across doses.
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 178 | 175
Subjects
  Any Fatigue, Dose 1: number analyzed (Participants) | 176 | 173
  Any Fatigue, Dose 1 | 30 | 39
  Grade 3 Fatigue, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 Fatigue, Dose 1 | 1 | 2
  Related Fatigue, Dose 1: number analyzed (Participants) | 176 | 173
  Related Fatigue, Dose 1 | 23 | 33
  Any GI symptoms, Dose 1: number analyzed (Participants) | 176 | 173
  Any GI symptoms, Dose 1 | 16 | 12
  Grade 3 GI symptoms, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 GI symptoms, Dose 1 | 1 | 1
  Related GI symptoms, Dose 1: number analyzed (Participants) | 176 | 173
  Related GI symptoms, Dose 1 | 9 | 5
  Any Headache, Dose 1: number analyzed (Participants) | 176 | 173
  Any Headache, Dose 1 | 21 | 20
  Grade 3 Headache, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 Headache, Dose 1 | 0 | 2
  Related Headache, Dose 1: number analyzed (Participants) | 176 | 173
  Related Headache, Dose 1 | 13 | 17
  Any Joint pain, Dose 1: number analyzed (Participants) | 176 | 173
  Any Joint pain, Dose 1 | 11 | 16
  Grade 3 Joint pain, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 Joint pain, Dose 1 | 0 | 0
  Related Joint pain, Dose 1: number analyzed (Participants) | 176 | 173
  Related Joint pain, Dose 1 | 6 | 14
  Any Muscle aches, Dose 1: number analyzed (Participants) | 176 | 173
  Any Muscle aches, Dose 1 | 15 | 20
  Grade 3 Muscle aches, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 Muscle aches, Dose 1 | 0 | 1
  Related Muscle aches, Dose 1: number analyzed (Participants) | 176 | 173
  Related Muscle aches, Dose 1 | 12 | 19
  Any Shivering, Dose 1: number analyzed (Participants) | 176 | 173
  Any Shivering, Dose 1 | 6 | 10
  Grade 3 Shivering, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 Shivering, Dose 1 | 0 | 1
  Related Shivering, Dose 1: number analyzed (Participants) | 176 | 173
  Related Shivering, Dose 1 | 5 | 8
  Any Sweating, Dose 1: number analyzed (Participants) | 176 | 173
  Any Sweating, Dose 1 | 11 | 16
  Grade 3 Sweating, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 Sweating, Dose 1 | 0 | 1
  Related Sweating, Dose 1: number analyzed (Participants) | 176 | 173
  Related Sweating, Dose 1 | 9 | 10
  Any Fever, Dose 1: number analyzed (Participants) | 176 | 173
  Any Fever, Dose 1 | 0 | 2
  Grade 3 Fever, Dose 1: number analyzed (Participants) | 176 | 173
  Grade 3 Fever, Dose 1 | 0 | 1
  Related Fever, Dose 1: number analyzed (Participants) | 176 | 173
  Related Fever, Dose 1 | 0 | 2
  Any Fatigue, Dose 2: number analyzed (Participants) | 177 | 171
  Any Fatigue, Dose 2 | 25 | 12
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 Fatigue, Dose 2 | 1 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 177 | 171
  Related Fatigue, Dose 2 | 22 | 6
  Any GI symptoms, Dose 2: number analyzed (Participants) | 177 | 171
  Any GI symptoms, Dose 2 | 11 | 7
  Grade 3 GI symptoms, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 GI symptoms, Dose 2 | 0 | 1
  Related GI symptoms, Dose 2: number analyzed (Participants) | 177 | 171
  Related GI symptoms, Dose 2 | 9 | 2
  Any Headache, Dose 2: number analyzed (Participants) | 177 | 171
  Any Headache, Dose 2 | 18 | 10
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 Headache, Dose 2 | 1 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 177 | 171
  Related Headache, Dose 2 | 14 | 3
  Any Joint pain, Dose 2: number analyzed (Participants) | 177 | 171
  Any Joint pain, Dose 2 | 17 | 11
  Grade 3 Joint pain, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 Joint pain, Dose 2 | 1 | 0
  Related Joint pain, Dose 2: number analyzed (Participants) | 177 | 171
  Related Joint pain, Dose 2 | 12 | 7
  Any Muscle aches, Dose 2: number analyzed (Participants) | 177 | 171
  Any Muscle aches, Dose 2 | 21 | 12
  Grade 3 Muscle aches, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 Muscle aches, Dose 2 | 4 | 0
  Related Muscle aches, Dose 2: number analyzed (Participants) | 177 | 171
  Related Muscle aches, Dose 2 | 19 | 6
  Any Shivering, Dose 2: number analyzed (Participants) | 177 | 171
  Any Shivering, Dose 2 | 8 | 5
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 Shivering, Dose 2 | 1 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 177 | 171
  Related Shivering, Dose 2 | 5 | 3
  Any Sweating, Dose 2: number analyzed (Participants) | 177 | 171
  Any Sweating, Dose 2 | 10 | 8
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 Sweating, Dose 2 | 1 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 177 | 171
  Related Sweating, Dose 2 | 5 | 5
  Any Fever, Dose 2: number analyzed (Participants) | 177 | 171
  Any Fever, Dose 2 | 1 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 177 | 171
  Grade 3 Fever, Dose 2 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 177 | 171
  Related Fever, Dose 2 | 1 | 0
  Any Fatigue, Across Doses | 43 | 43
  Grade 3 Fatigue, Across Doses | 2 | 2
  Related Fatigue, Across Doses | 34 | 37
  Any GI symptoms, Across Doses | 23 | 17
  Grade 3 GI symptoms, Across Doses | 1 | 2
  Related GI symptoms, Across Doses | 15 | 7
  Any Headache, Across Doses | 30 | 27
  Grade 3 Headache, Across Doses | 1 | 2
  Related Headache, Across Doses | 22 | 20
  Any Joint pain, Across Doses | 25 | 23
  Grade 3 Joint pain, Across Doses | 1 | 0
  Related Joint pain, Across Doses | 16 | 20
  Any Muscle aches, Across Doses | 32 | 28
  Grade 3 Muscle aches, Across Doses | 4 | 1
  Related Muscle aches, Across Doses | 28 | 24
  Any Shivering, Across Doses | 13 | 14
  Grade 3 Shivering, Across Doses | 1 | 1
  Related Shivering, Across Doses | 9 | 10
  Any Sweating, Across Doses | 16 | 19
  Grade 3 Sweating, Across Doses | 1 | 1
  Related Sweating, Across Doses | 11 | 14
  Any Fever, Across Doses | 1 | 2
  Grade 3 Fever, Across Doses | 0 | 1
  Related Fever, Across Doses | 1 | 2

5. Secondary Outcome: Duration of Local Adverse Events
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 63 | 90
Days
  Pain, Dose 1: number analyzed (Participants) | 35 | 90
  Pain, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Pain, Dose 2: number analyzed (Participants) | 63 | 8
  Pain, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Redness, Dose 1: number analyzed (Participants) | 6 | 9
  Redness, Dose 1 | 4.0 [3.0 to 4.0] | 2.0 [2.0 to 3.0]
  Redness, Dose 2: number analyzed (Participants) | 8 | 1
  Redness, Dose 2 | 2.0 [1.0 to 2.5] | 1.0 [1.0 to 1.0]
  Swelling, Dose 1: number analyzed (Participants) | 2 | 9
  Swelling, Dose 1 | 4.5 [4.0 to 5.0] | 2.0 [2.0 to 4.0]
  Swelling, Dose 2: number analyzed (Participants) | 5 | 0
  Swelling, Dose 2 | 3.0 [1.0 to 5.0] |

6. Secondary Outcome: Duration of Solicited General AEs.
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period
Population: as for outcome 3
Measure: Median (Full Range); unit: Days
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 30 | 39
Days
  Fatigue, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Fatigue, Dose 2: number analyzed (Participants) | 25 | 12
  Fatigue, Dose 2 | 3.0 [2.0 to 4.0] | 3.5 [1.5 to 6.5]
  Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 16 | 12
  Gastrointestinal symptoms, Dose 1 | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 2.0]
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 11 | 7
  Gastrointestinal symptoms, Dose 2 | 3.0 [2.0 to 3.0] | 3.0 [2.0 to 6.0]
  Headache, Dose 1: number analyzed (Participants) | 21 | 20
  Headache, Dose 1 | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 2.5]
  Headache, Dose 2: number analyzed (Participants) | 18 | 10
  Headache, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Joint pain, Dose 1: number analyzed (Participants) | 11 | 16
  Joint pain, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Joint pain, Dose 2: number analyzed (Participants) | 17 | 11
  Joint pain, Dose 2 | 2.0 [2.0 to 3.0] | 2.0 [1.0 to 7.0]
  Muscle aches, Dose 1: number analyzed (Participants) | 15 | 20
  Muscle aches, Dose 1 | 2.0 [1.0 to 3.0] | 3.0 [1.5 to 4.5]
  Muscle aches, Dose 2: number analyzed (Participants) | 21 | 12
  Muscle aches, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Sweating, Dose 1: number analyzed (Participants) | 11 | 16
  Sweating, Dose 1 | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 3.5]
  Sweating, Dose 2: number analyzed (Participants) | 10 | 8
  Sweating, Dose 2 | 2.0 [1.0 to 5.0] | 2.0 [1.5 to 2.0]
  Shivering, Dose 1: number analyzed (Participants) | 6 | 10
  Shivering, Dose 1 | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Shivering, Dose 2: number analyzed (Participants) | 8 | 5
  Shivering, Dose 2 | 1.0 [1.0 to 2.0] | 3.0 [1.0 to 3.0]
  Fever, Dose 1: number analyzed (Participants) | 0 | 2
  Fever, Dose 1 |  | 1.0 [1.0 to 1.0]
  Fever, Dose 2: number analyzed (Participants) | 1 | 0
  Fever, Dose 2 | 1.0 [1.0 to 1.0] |

7. Secondary Outcome: Number of Subjects Reporting the Occurrence of Medically Attended Adverse Events (MAEs)
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s) regardless of intensity grade or relationship to vaccination. Related was defined as MAE assessed by the investigator to be causally related to the study vaccination.
Time Frame: Throughout the study period (Days 0-180)
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 179 | 177
Subjects
  Any MAE(s) | 37 | 43
  Related MAE(s) | 2 | 2

8. Secondary Outcome: Number of Subjects Reporting the Occurrence of Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) were defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
  Any was defined as any occurrence of pIMD(s) regardless of intensity grade or relationship to vaccination. Related was defined as pIMD assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the entire study period (Days 0-180)
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 179 | 177
Subjects
  Any pIMD(s) | 0 | 1
  Related pIMD(s) | 0 | 0

9. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination.
Time Frame: Within the 28-day (Days 0-27) post-vaccination period
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 179 | 177
Subjects
  Any Unsolicited AEs | 35 | 42
  Grade 3 Unsolicited AEs | 5 | 8
  Related Unsolicited AEs | 5 | 5

10. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Throughout the study period (Days 0-180)
Population: as for outcome 3
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 179 | 177
Subjects
  Any SAE(s) | 11 | 7
  Related SAE(s) | 0 | 0
  Fatal SAE(s) | 0 | 1
  Related Fatal SAE(s) | 0 | 0

11. Secondary Outcome: Humoral Immune Response in Terms of Haemagglutination Inhibition (HI) Antibodies in Subjects by Calculating Serum Antihaemagglutination (HA) Antibody Titers Against the 4 Influenza Vaccine Strains
Description: HI antibody titres were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Brisbane/60/2008 (Victoria) and Flu B/Massachusetts/02/2012 (Yamagata).
Time Frame: At Day 0 and Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 171 | 163
Titers
  H1N1, Day 0: number analyzed (Participants) | 171 | 162
  H1N1, Day 0 | 32.4 [26.3 to 39.9] | 253.2 [205.3 to 312.1]
  H1N1, Day 28: number analyzed (Participants) | 170 | 163
  H1N1, Day 28 | 34.0 [27.8 to 41.7] | 235.5 [195.0 to 284.5]
  H3N2, Day 0: number analyzed (Participants) | 171 | 162
  H3N2, Day 0 | 20.8 [17.5 to 24.9] | 21.8 [18.2 to 26.2]
  H3N2, Day 28: number analyzed (Participants) | 170 | 162
  H3N2, Day 28 | 73.6 [62.1 to 87.1] | 78.6 [65.2 to 94.7]
  Victoria, Day 0: number analyzed (Participants) | 171 | 162
  Victoria, Day 0 | 48.7 [41.6 to 57.1] | 51.5 [43.9 to 60.3]
  Victoria, Day 28: number analyzed (Participants) | 170 | 162
  Victoria, Day 28 | 178.7 [154.9 to 206.2] | 157.9 [136.4 to 182.9]
  Yamagata, Day 0: number analyzed (Participants) | 171 | 162
  Yamagata, Day 0 | 120.7 [104.3 to 139.8] | 119.9 [103.0 to 139.5]
  Yamagata, Day 28: number analyzed (Participants) | 170 | 162
  Yamagata, Day 28 | 346.5 [302.3 to 397.1] | 353.8 [310.5 to 403.2]

12. Secondary Outcome: Number of Subjects Who Were Seroprotected for Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Brisbane/60/2008 (Victoria) and Flu B/Massachusetts/2/2012 (Yamagata).
Time Frame: At Day 0 and Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 171 | 163
Subjects
  H1N1, Day 0: number analyzed (Participants) | 171 | 162
  H1N1, Day 0 | 83 | 77
  H1N1, Day 28: number analyzed (Participants) | 170 | 163
  H1N1, Day 28 | 160 | 157
  H3N2, Day 0: number analyzed (Participants) | 171 | 162
  H3N2, Day 0 | 57 | 50
  H3N2, Day 28: number analyzed (Participants) | 170 | 162
  H3N2, Day 28 | 131 | 128
  Victoria, Day 0: number analyzed (Participants) | 171 | 162
  Victoria, Day 0 | 106 | 113
  Victoria, Day 28: number analyzed (Participants) | 170 | 162
  Victoria, Day 28 | 167 | 154
  Yamagata, Day 0: number analyzed (Participants) | 171 | 162
  Yamagata, Day 0 | 159 | 146
  Yamagata, Day 28: number analyzed (Participants) | 170 | 162
  Yamagata, Day 28 | 169 | 162

13. Secondary Outcome: Number of Seroconverted Subjects for Anti-Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Brisbane/60/2008 (Victoria) and Flu B/Massachusetts/02/2012 (Yamagata).
Time Frame: At Day 28
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 170 | 162
Subjects
  H1N1 | 110 | 101
  H3N2 | 62 | 61
  Victoria | 73 | 55
  Yamagata | 60 | 54

14. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the Four Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum haemagglutination inhibition (HI) GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/Christchurch/16/2010 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Brisbane/60/2008 (Victoria) and Flu B/Massachusetts/02/2012 (Yamagata).
Time Frame: At Day 28
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 170 | 162
Fold increase
  H1N1 | 7.7 [6.1 to 9.7] | 6.9 [5.5 to 8.6]
  H3N2 | 3.5 [3.0 to 4.2] | 3.6 [3.0 to 4.4]
  Victoria | 3.6 [3.1 to 4.3] | 3.1 [2.6 to 3.6]
  Yamagata | 2.8 [2.5 to 3.3] | 3.0 [2.5 to 3.4]

15. Secondary Outcome: Number of Subjects With Anti-pneumococcal Antibody Concentrations for the Following Serotypes: 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F
Description: The pneumococcal antigen testing was performed, as determined by ELISA cut-offs of ≥0.05 µg/mL and a seroprotection cut-off of ≥ 0.2 µg/ml.
  PRE = Pre-vaccination i.e. at Day 0 for Co-Ad Group and at Day 28 for Control Group.
  POST = Post-vaccination i.e. at Day 28 for Co-Ad Group and at Day 56 for Control Group.
Time Frame: At Days 0 (Co-Ad group only), 28 (both groups), and 56 (Control group only)
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 170 | 163
Subjects
  Polysaccharide 01 Ab.IgG (≥ 0.05 µg/ml) (PRE) | 162 | 152
  Polysaccharide 01 Ab.IgG (≥ 0.05 µg/ml) (POST) | 169 | 162
  Polysaccharide 01 Ab.IgG (≥ 0.2 µg/ml) (PRE) | 112 | 118
  Polysaccharide 01 Ab.IgG (≥ 0.2 µg/ml) (POST) | 167 | 159
  Polysaccharide 03 Ab.IgG (≥ 0.05 µg/ml) (PRE) | 158 | 149
  Polysaccharide 03 Ab.IgG (≥ 0.05 µg/ml) (POST) | 167 | 161
  Polysaccharide 03 Ab.IgG (≥ 0.2 µg/ml) (PRE) | 114 | 121
  Polysaccharide 03 Ab.IgG (≥ 0.2 µg/ml) (POST) | 158 | 153
  Polysaccharide 04 Ab.IgG (≥ 0.05 µg/ml) (PRE) | 138 | 129
  Polysaccharide 04 Ab.IgG (≥ 0.05 µg/ml) (POST) | 167 | 158
  Polysaccharide 04 Ab.IgG (≥ 0.2 µg/ml) (PRE) | 77 | 82
  Polysaccharide 04 Ab.IgG (≥ 0.2 µg/ml) (POST) | 158 | 149
  Polysaccharide 05 Ab.IgG5 (≥ 0.05 µg/ml) (PRE) | 165 | 159
  Polysaccharide 05 Ab.IgG5 (≥ 0.05 µg/ml) (POST) | 169 | 162
  Polysaccharide 05 Ab.IgG5 (≥ 0.2 µg/ml) (PRE) | 130 | 115
  Polysaccharide 05 Ab.IgG5 (≥ 0.2 µg/ml) (POST) | 163 | 155
  Polysaccharide 6B Ab.IgG (≥ 0.05 µg/ml) (PRE) | 158 | 149
  Polysaccharide 6B Ab.IgG (≥ 0.05 µg/ml) (POST) | 164 | 160
  Polysaccharide 6B Ab.IgG (≥ 0.2 µg/ml) (PRE) | 106 | 110
  Polysaccharide 6B Ab.IgG (≥ 0.2 µg/ml) (POST) | 157 | 147
  Polysaccharide 7F Ab.IgG (≥ 0.05 µg/ml) (PRE) | 159 | 154
  Polysaccharide 7F Ab.IgG (≥ 0.05 µg/ml) (POST) | 169 | 162
  Polysaccharide 7F Ab.IgG (≥ 0.2 µg/ml) (PRE) | 127 | 130
  Polysaccharide 7F Ab.IgG (≥ 0.2 µg/ml) (POST) | 165 | 161
  Polysaccharide 9V Ab.IgG (≥ 0.05 µg/ml) (PRE) | 165 | 150
  Polysaccharide 9V Ab.IgG (≥ 0.05 µg/ml) (POST) | 168 | 160
  Polysaccharide 9V Ab.IgG (≥ 0.2 µg/ml) (PRE) | 123 | 117
  Polysaccharide 9V Ab.IgG (≥ 0.2 µg/ml) (POST) | 166 | 157
  Polysaccharide 14 Ab.IgG (≥ 0.05 µg/ml) (PRE) | 170 | 163
  Polysaccharide 14 Ab.IgG (≥ 0.05 µg/ml) (POST) | 169 | 162
  Polysaccharide 14 Ab.IgG (≥ 0.2 µg/ml) (PRE) | 168 | 160
  Polysaccharide 14 Ab.IgG (≥ 0.2 µg/ml) (POST) | 168 | 162
  Polysaccharide 18C Ab.IgG (≥ 0.05 µg/ml) (PRE) | 166 | 161
  Polysaccharide 18C Ab.IgG (≥ 0.05 µg/ml) (POST) | 169 | 162
  Polysaccharide 18C Ab.IgG (≥ 0.2 µg/ml) (PRE) | 154 | 148
  Polysaccharide 18C Ab.IgG (≥ 0.2 µg/ml) (POST) | 168 | 159
  Polysaccharide 19A Ab.IgG (≥ 0.05 µg/ml) (PRE) | 168 | 160
  Polysaccharide 19A Ab.IgG (≥ 0.05 µg/ml) (POST) | 169 | 161
  Polysaccharide 19A Ab.IgG (≥ 0.2 µg/ml) (PRE) | 146 | 148
  Polysaccharide 19A Ab.IgG (≥ 0.2 µg/ml) (POST) | 165 | 158
  Polysaccharide 19F Ab.IgG (≥ 0.05 µg/ml) (PRE) | 169 | 160
  Polysaccharide 19F Ab.IgG (≥ 0.05 µg/ml) (POST) | 169 | 162
  Polysaccharide 19F Ab.IgG (≥ 0.2 µg/ml) (PRE) | 151 | 152
  Polysaccharide 19F Ab.IgG (≥ 0.2 µg/ml) (POST) | 169 | 161
  Polysaccharide 23F Ab.IgG (≥ 0.05 µg/ml) (PRE) | 151 | 151
  Polysaccharide 23F Ab.IgG (≥ 0.05 µg/ml) (POST) | 165 | 159
  Polysaccharide 23F Ab.IgG (≥ 0.2 µg/ml) (PRE) | 112 | 125
  Polysaccharide 23F Ab.IgG (≥ 0.2 µg/ml) (POST) | 155 | 147

16. Secondary Outcome: Pneumococcal Vaccine Response in Terms of Anti-pneumococcal Antibody Concentrations Against 12 Pneumococcal Serotypes (1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F)
Description: Anti-pneumococcal antibody concentrations were expressed as adjusted geometric mean concentrations (GMCs) PRE = Pre -vaccination i.e. at Day 0 for Co-Ad Group and at Day 28 for Control Group.
  POST = Post-vaccination i.e. at Day 28 for Co-Ad Group and at Day 56 for Control Group.
Time Frame: At Days 0 (Co-Ad group only), 28 (both groups), and 56 (Control group only)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 170 | 163
Titers
  Polysaccharide 01 Ab.IgG (PRE) | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.5]
  Polysaccharide 01 Ab.IgG (POST) | 5.5 [4.3 to 7.0] | 4.9 [3.9 to 6.2]
  Polysaccharide 03 Ab.IgG (PRE) | 0.4 [0.3 to 0.5] | 0.5 [0.4 to 0.6]
  Polysaccharide 03 Ab.IgG (POST) | 1.7 [1.4 to 2.1] | 1.7 [1.4 to 2.0]
  Polysaccharide 04 Ab.IgG (PRE) | 0.2 [0.2 to 0.3] | 0.2 [0.2 to 0.2]
  Polysaccharide 04 Ab.IgG (POST) | 2.3 [1.8 to 2.9] | 1.7 [1.4 to 2.2]
  Polysaccharide 05 Ab.IgG5 (PRE) | 0.6 [0.5 to 0.7] | 0.5 [0.4 to 0.6]
  Polysaccharide 05 Ab.IgG5 (POST) | 7.8 [5.9 to 10.4] | 5.7 [4.3 to 7.5]
  Polysaccharide 6B Ab.IgG (PRE) | 0.4 [0.3 to 0.6] | 0.4 [0.3 to 0.5]
  Polysaccharide 6B Ab.IgG (POST) | 3.9 [2.9 to 5.1] | 3.1 [2.3 to 4.1]
  Polysaccharide 7F Ab.IgG (PRE) | 0.6 [0.5 to 0.8] | 0.7 [0.6 to 0.9]
  Polysaccharide 7F Ab.IgG (POST) | 9.0 [6.9 to 11.8] | 8.1 [6.2 to 10.6]
  Polysaccharide 9V Ab.IgG (PRE) | 0.5 [0.4 to 0.7] | 0.5 [0.4 to 0.6]
  Polysaccharide 9V Ab.IgG (POST) | 5.9 [4.8 to 7.4] | 4.4 [3.6 to 5.5]
  Polysaccharide 14 Ab.IgG (PRE) | 3.7 [3.1 to 4.6] | 2.9 [2.4 to 3.5]
  Polysaccharide 14 Ab.IgG (POST) | 20.2 [16.0 to 25.6] | 14.1 [11.3 to 17.6]
  Polysaccharide 18C Ab.IgG (PRE) | 1.4 [1.1 to 1.7] | 1.2 [1.0 to 1.5]
  Polysaccharide 18C Ab.IgG (POST) | 13.5 [10.7 to 16.8] | 11.1 [9.0 to 13.6]
  Polysaccharide 19A Ab.IgG (PRE) | 1.3 [1.0 to 1.6] | 1.5 [1.2 to 1.9]
  Polysaccharide 19A Ab.IgG (POST) | 9.2 [7.1 to 11.9] | 7.7 [6.1 to 9.8]
  Polysaccharide 19F Ab.IgG (PRE) | 1.3 [1.1 to 1.7] | 1.4 [1.2 to 1.8]
  Polysaccharide 19F Ab.IgG (POST) | 11.9 [9.3 to 15.2] | 10.6 [8.4 to 13.6]
  Polysaccharide 23F Ab.IgG (PRE) | 0.4 [0.3 to 0.6] | 0.5 [0.4 to 0.7]
  Polysaccharide 23F Ab.IgG (POST) | 3.1 [2.3 to 4.1] | 2.9 [2.2 to 3.8]

17. Secondary Outcome: Number of Subjects Whose N Antibody Titers Were at Least 2 or 4-fold Higher Than Their Pre-vaccination Titer by Anti-pneumococcal Serotype Subjects.
Description: Fold antibody concentration increases post-vaccination/pre-vaccination ≥ 2 and ≥ 4.
  The anti-pneumococcal serotypes assessed were 1, 3, 4, 5, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F.
Time Frame: At 28 days post-vaccination with Pneumovax™ 23
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Control Group | Co-Ad Group
Number analyzed (Participants) | 169 | 163
Subjects
  Polysaccharide 01 Ab.IgG (≥ 2) | 149 | 144
  Polysaccharide 01 Ab.IgG (≥ 4) | 134 | 126
  Polysaccharide 03 Ab.IgG (≥ 2) | 121 | 97
  Polysaccharide 03 Ab.IgG (≥ 4) | 80 | 65
  Polysaccharide 04 Ab.IgG (≥ 2) | 149 | 137
  Polysaccharide 04 Ab.IgG (≥ 4) | 127 | 112
  Polysaccharide 05 Ab.IgG5 (≥ 2) | 156 | 138
  Polysaccharide 05 Ab.IgG5 (≥ 4) | 127 | 114
  Polysaccharide 14 Ab.IgG (≥ 2) | 123 | 102
  Polysaccharide 14 Ab.IgG (≥ 4) | 90 | 82
  Polysaccharide 18C Ab.IgG (≥ 2) | 149 | 133
  Polysaccharide 18C Ab.IgG (≥ 4) | 123 | 116
  Polysaccharide 19A Ab.IgG (≥ 2) | 133 | 123
  Polysaccharide 19A Ab.IgG (≥ 4) | 111 | 87
  Polysaccharide 19F Ab.IgG (≥ 2) | 146 | 141
  Polysaccharide 19F Ab.IgG (≥ 4) | 111 | 109
  Polysaccharide 23F Ab.IgG (≥ 2) | 133 | 122
  Polysaccharide 23F Ab.IgG (≥ 4) | 108 | 94
  Polysaccharide 6B Ab.IgG (≥ 2) | 141 | 127
  Polysaccharide 6B Ab.IgG (≥ 4) | 113 | 109
  Polysaccharide 7F Ab.IgG (≥ 2) | 155 | 144
  Polysaccharide 7F Ab.IgG (≥ 4) | 138 | 119
  Polysaccharide 9V Ab.IgG (≥ 2) | 146 | 140
  Polysaccharide 9V Ab.IgG (≥ 4) | 131 | 121

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: During the entire study period (Day 0 to 180); Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events: During the 28-day (Days 0-27) post-vaccination period.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated cohort who had the symptom sheet completed.
Arm/Group | Control Group | Co-Ad Group
Serious Adverse Events (participants affected / at risk) | 11/179 | 7/177
Other Adverse Events (participants affected / at risk) | 117/179 | 127/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=179) | Co-Ad Group (N=177)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal malrotation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Calcinosis (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cancer stage ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=179) | Co-Ad Group (N=177)
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (28) | 25 (30)
Chills (General disorders) | 13 (14) | 14 (15)
Erythema (Skin and subcutaneous tissue disorders) | 13 (14) | 10 (10)
Fatigue (General disorders) | 43 (55) | 43 (51)
Gastrointestinal disorder (Gastrointestinal disorders) | 23 (27) | 17 (19)
Headache (Nervous system disorders) | 31 (41) | 27 (30)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 16 (21) | 19 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 32 (36) | 28 (32)
Pain (General disorders) | 76 (98) | 92 (98)
Swelling (General disorders) | 6 (7) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.